CLINICAL TRIAL: NCT06780202
Title: Assessment of Medrol Dosepak to Reduce Opioid Consumption in Foot and Ankle Surgical Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jason Bariteau, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008454
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Foot Injuries and Disorders; Ankle Injuries and Disorders; Achilles Tendon Injury
Keywords: VAS scale: visual analog scale; Medrol Dosepak
MeSH Terms: conditions — Foot Injuries; Disease; Ankle Injuries | interventions — Methylprednisolone; Hydrocodone

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medrol (Experimental): The group will be given Medrol Dosepak in a tapered, low-dose manner, orally once a day.
  Subjects will be sent home with a pain journal where they will record their pain and nausea 3 times daily starting the day of surgery and the following 7 days along with their daily hydrocodone consumption. These journals will be collected at their 2-week post-op appointment which is scheduled ± 1 week. In this appointment, subjects will also be evaluated for complications.
  Interventions: Drug: medrol dosepak; Drug: HYDROcodone Oral Tablet
- Standard of Care (Active Comparator): Each subject will receive the standard pain regime of both surgeons. This includes a nerve block before surgery for pain prevention. While in surgery, the subject will receive 10 mg of dexamethasone intravenously. Post-surgery, each subject will be instructed to take vitamin C for nerve pain and vitamin D for bone healing. They will also be provided with a prescription of aspirin for deep vein thrombosis (DVT) prophylaxis, ondansetron (Zofran) for nausea, and Colace for constipation relief. Both groups will receive a prescription of 20 5 mg hydrocodone pills to be taken as needed for pain, 1 every 6 hours
  Subjects will be sent home with a pain journal where they will record their pain and nausea 3 times starting the day of surgery and the following 7 days along with their daily hydrocodone consumption. Journals will be collected at their 2-week post-op appointment which is scheduled ± 1 week. Subjects will also be evaluated for complications
  Interventions: Drug: HYDROcodone Oral Tablet

INTERVENTIONS:
Drug: medrol dosepak — Methylprednisolone is a corticosteroid with anti-inflammatory properties and immune suppression.
  This study will utilize a 6-day Medrol Dosepak: a tapered low-dose corticosteroid course taken orally once a day. This includes 6 tablets on day 1 (24 mg), 5 tablets on day 2 (20 mg), 4 tablets on day 3 (16 mg), 3 tablets on day 4 (12 mg), 2 tablets on day 5 (8 mg) and 1 tablet on day 6 (4 mg).
  Other Names: Methylprednisolone
  Arms: Medrol
Drug: HYDROcodone Oral Tablet — This study will utilize a prescription of 20 pills of hydrocodone, 5mg each, to be taken as needed for pain, 1 every 6 hours.

SUMMARY:
This clinical trial aims to determine the effects of a 6-day low-dose methylprednisolone course on pain, nausea, and total opioid consumption in patients undergoing foot and ankle surgeries.

The secondary objective of the study is to determine and monitor the effects of the course on complications following surgery and patient-reported outcomes

DETAILED DESCRIPTION:
The opioid epidemic continues to create a lasting impact on society, leading researchers to focus on ways to decrease opioid prescription rates and subsequently, opioid consumption. Opioid-naïve patients undergoing minor to major surgeries have been shown statistically to be largely affected.1 This includes significant numbers resulting from forefoot surgery specifically with around 6.2% of the mentioned population being at risk for new persistent opioid use.

This has provoked researchers to seek a new route that decreases exposure to opioid use through proposals for multimodal pain regimes.

A recent addition to some of these proposed treatments has been a 6-day low-dose oral methylprednisolone taper beginning on the day of surgery. This has been tested with "terrible triad" elbow injuries, distal radius fractures, and total shoulder arthroplasties with promising results showing decreased consumption of the as-needed opioid prescription. Furthermore, the results of these studies show a significant decrease in pain and increased range of motion following surgery. This is likely due to the anti-inflammatory functioning of glucocorticoids, without inhibiting the healing process.

Based upon the findings stated above, the proposed research will attempt to apply this new pain regime to foot and ankle surgeries, specifically forefoot, ankle, and Achilles surgeries, to take another step towards bettering perioperative care with opioid-free treatment

ELIGIBILITY:
Inclusion Criteria:

-Emory Orthopedic patients undergoing foot and ankle surgery

Exclusion Criteria:

* Concurrent or significant injuries to other bones or organs
* Local infections
* History of alcohol or medical abuse, including prior opioid abuse
* Smoking
* History of severe heart disease, renal failure, liver dysfunction, active peptic ulcer disease, diabetes, rheumatoid arthritis, neurological or psychiatric diseases that could influence pain perception
* Pre-existing immune suppression
* Those deemed possibly non-compliant by the study team and,
* All vulnerable populations (those unable to give consent, juveniles, pregnant women, prisoners, cognitively impaired and non-English speaking).

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post operative Nausea | Baseline (Day 0), 7 days post op
  The subjects will report nausea along the visual analog scale (VAS scale), which they will be educated on before surgery.
  A VAS for nausea is a straight line with one end labeled "no nausea" and the other end labeled "worst nausea imaginable". The patient marks a point on the line to indicate their nausea level. The distance from the "no nausea" end of the line is used to score the nausea intensity
Post operative pain | Baseline, 0.25 months, 1.5 months, 3 months, 6 months
  The subject will measure pain along the visual analog scale (VAS scale), which they will be educated on before surgery.
  A VAS for pain is a straight line with one end labeled "no pain" and the other end labeled "worst pain imaginable". The patient marks a point on the line to indicate their pain level. The distance from the "no pain" end of the line is used to score the pain intensity
Post operative opioid consumption | Baseline (Day 0), 7 days post op
  Total number of opioids consumed each day will be captured.

SECONDARY OUTCOMES:
Complications due to the Medrol Dosepak | 1.5 months, 3 months, 6 months
  Complications will be monitored via radiographs and clinical analyses at post-operative appointments for impaired wound-healing and infection
Patient reported outcomes | Baseline (pre operative assessment), Post operation (6 months)
  Patient-reported outcomes will be measured along the 12-item Short Form Health Survey which measures the impact of their current health on everyday life, the Patient-Reported Outcomes Measurement Information System (PROMIS) which measures physical, mental, and social health and the VAS scale, which measures pain at rest

CONTACTS AND LOCATIONS:
Overall Officials: Rishin Kadakia, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Musculoskeletal Institute, Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Emory Sports Medicine Complex and Emory Orthopaedics and Spine Center, Johns Creek, Georgia